CLINICAL TRIAL: NCT02695875
Title: Comparative Study About the Effect of a Physical Therapy Protocol in Warm Water vs Land-based Therapy in Women With Fibromyalgia Syndrome
Brief Title: Comparative Study About the Effect of Aquatic Therapy vs Land-based Therapy in Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Sabela Rivas Neira, PhD, PhD, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIB-2014
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain; Postural balance; Physical therapy; Aquatic therapy
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aquatic therapy (Experimental): Aquatic therapy is the experimental group. This therapy will take place in a warm pool which is located in Rialta's Sports Complex. Aquatic therapy session will be conducted by the main researcher with the help of an assistant. Because the number of patients (n=17), they will be subdivided into two subgroups of 8 and 9 people respectively in order to ensure the safety and care of patients. The intervention will last for one hour: Warming (15 minutes); exercises to train the static and dynamic balance (25 minutes); stretching (10 minutes); relaxation (10 minutes). Over 12 weeks of treatment, difficulty in performing exercises to train balance will increase progressively.
  Interventions: Procedure: Aquatic therapy
- Land-based therapy (Other): The description is the same as aquatic therapy. The difference is land-based therapy sessions will be made at Faculty of Physiotherapy at University of "A Coruña".
  Interventions: Procedure: Land-based therapy

INTERVENTIONS:
Procedure: Aquatic therapy — Pool material is contributed by Maria José Jove Foundation. The exercises that will be made during treatment, are designed and developed to improve "core" muscles and, in this way, improve postural balance.
  Arms: Aquatic therapy
Procedure: Land-based therapy — The material is contributed by Faculty of Physiotherapy at University of "A Coruña".
  The exercises that will be made during treatment, are designed and developed to improve "core" muscles and, in this way, improve postural balance.
  Arms: Land-based therapy

SUMMARY:
Fibromyalgia is a disease whose incidence rate is increasing and causing a severe disability to those who suffer it. Currently, other treatment resources are being implemented, such as aquatic therapy. This therapy seems to provide positive results in different dimensions of fibromyalgia.

The main objective of the study is to determine the effectiveness of a physical therapy program in warm water vs. land-based therapy in women with fibromyalgia for pain reduction and improvement balance at the end of treatment and a month and a half later (follow-up).

The type of study is a randomized controlled opened trial. The sample is composed of 34 women with age between 35 and 64 years and fibromyalgia diagnosis who will be divided into 2 groups: Aquatic Therapy Group (n=17) and Land-Based Therapy Group (n=17). This study will have two primary outcomes: Pain and balance. The intensity of pain will be assessed using the visual analog scale (VAS) and the pain threshold for each one of the 18 tender points will be assessed using a electronic algometer. Static balance will be evaluated with the Romberg's test and the dynamic balance with the Timed Up & Go test (TUG) and Berg Balance Scale. Both type of balance will be recorded in slow motion and then, will be analysed with a motion software. Secondary outcomes are: The impact of fibromyalgia on patient's lives, that will be measured with the "Revised Fibromyalgia Impact Questionnaire" (FIQR); the sleep quality, that will be assessed with the "Pittsburgh Sleep Quality Index" (PSQI); the fatigue, that will be evaluated witn the "Multidimensional Fatigue Inventory" (MFI); the physical capacity, that will be measured with the "six minute walk test" (SMWT) and confidence in balance that will be assessed with the "Activities-specific Balance Confidence" scale (ABC).

Each intervention will last one hour and will be made 3 times a week for three months . It will consist of 4 sections: Warming, exercises for static and dynamic balance training, stretching and relaxation. Statistical analysis will be made using the Statistical Package for the Social Sciences software, version 21.0 for Windows. p ≤ 0.05 will be the significance level set for all analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Age range between 35 and 64 years.
* Diagnosis of fibromyalgia according to the criteria of the American College of Rheumatology (ACR) in 1990 and 2010.
* Mark ≥ 4 on the Visual Analogue Scale (VAS).
* Mark ≥ 5 on the Visual Analogue Scale for balance included in The Revised Fibromyalgia Impact Questionnaire (FIQR).

Exclusion Criteria:

* History of severe trauma.
* Neurological diseases (stroke, Parkinson's disease, dementia).
* Frequent migraines.
* Inflammatory rheumatic diseases.
* People who have been treated in the past six months by traumatic injuries.
* Being pregnant.
* Visual or hearing deficits uncorrected.
* Infectious diseases.
* Severe cardiovascular disease.
* People who do exercise regularly more than 20 minutes, more than 3 times a week in the past 3 months.

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Pain at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  Pain will be assessed using the visual analog scale (VAS).
Change from baseline Static Balance at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  It will be evaluated with the Romberg's test, whose execution will be filmed in slow motion and then, these videos will be analysed with a motion software.
Change from baseline Dynamic Balance at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  It will be assessed using the Timed Up & Go test (TUG), whose execution will be filmed in slow motion and then, these videos will be analysed with a motion software.

SECONDARY OUTCOMES:
Change from baseline Quality of Life at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  It will be measured with the "Revised Fibromyalgia Impact Questionnaire" (FIQR).
Change from baseline Sleep Quality at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  It will be assessed with the "Pittsburgh Sleep Quality Index" (PSQI).
Change from baseline Fatigue at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  It will be evaluated with the "Multidimensional Fatigue Inventory" (MFI).
Change from baseline Physical Capacity at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  It will be measured with the "six minute walk test" (SMWT).
Change from baseline Confidence in Balance at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  It will be assessed with the "Activities-specific Balance Confidence" scale (ABC).
Change from baseline Pain Threshold for each one of the 18 tender points established at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  It will be assessed using an electronic algometer.
Change from baseline Functional Independence to perform activities of daily living at 3 months of therapy and one month and a half after treatment. | It will be measured at baseline, at 3 months of therapy and one month and a half after treatment (follow-up).
  It will be assessed using the Berg Balance Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sabela Rivas Neira, Physiotherapy, Principal Investigator — Facultade de Fisioterapia da Universidade da Coruña; Jamile Vivas Costa, Physiotherapy, Study Director — Facultade de Fisioterapia da Universidade da Coruña
Locations (1):
- Asociación Coruñesa de Fibromialgia, Síndrome de Fatiga Crónica y Sensibilidad Química Múltiple (ACOFIFA), A Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rivas Neira S, Pasqual Marques A, Fernandez Cervantes R, Seoane Pillado MT, Vivas Costa J. Efficacy of aquatic vs land-based therapy for pain management in women with fibromyalgia: a randomised controlled trial. Physiotherapy. 2024 Jun;123:91-101. doi: 10.1016/j.physio.2024.02.005. Epub 2024 Feb 17. PMID 38447497
- [Derived] Rivas Neira S, Pasqual Marques A, Pegito Perez I, Fernandez Cervantes R, Vivas Costa J. Effectiveness of Aquatic Therapy vs Land-based Therapy for Balance and Pain in Women with Fibromyalgia: a study protocol for a randomised controlled trial. BMC Musculoskelet Disord. 2017 Jan 19;18(1):22. doi: 10.1186/s12891-016-1364-5. PMID 28103853